CLINICAL TRIAL: NCT06689410
Title: Multimodal Biocollection Linked to the French Register of Intracranial Aneurysms
Acronym: bCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Federation of Medical Specialties (Other); Inserm UMR1087, CNRS UMR6291 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC24_0512
Record Dates: First submitted 2024-10-31; First posted 2024-11-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-11

CONDITIONS: Aneurysm; Brain Aneurysm; Congenital Disease
Keywords: intracranial aneurysm; phenotype; genetics; imaging; multimodal data
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm; Congenital, Hereditary, and Neonatal Diseases and Abnormalities | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICA cases (Other): Any adult patient consulting for a definite and typical bifurcation AIC authenticated on MRI and/or cerebral arteriography
  Interventions: Other: blood or saliva sample

INTERVENTIONS:
Other: blood or saliva sample — Collection of blood or saliva

SUMMARY:
The purpose of the bCAN study is to create a prospective collection of multimodal data and human samples, linked to the French Intracranial Aneurysm Registry (FRAN).

The aim of bCAN is to enable risk stratification of ruptured ICAs by redefining "intracranial aneurysm disease". The description of genotypically and phenotypically specific subgroups of cases will pave the way for improved patient management based on new diagnostic/prognostic strategies among AIC carriers, either in a familial context, or at the level of the general population.

DETAILED DESCRIPTION:
The main objective of bCAN study is to build a predictive model of intracranial aneurysm phenotypes through the combination of information on genetic mutations, imaging findings and ICA rupture characteristics.

The secondary objectives of the bCAN study are (i) to study morphological characterization of ICA and vascular bifurcations, (ii) to deepen knowledge of genotype/clinical and biological phenotype relationships according to the genes identified in the different families, (iii) to research and validate the relationships between genotypes and phenotypes (including rupture) of ICA in a large population of sporadic ICA cases.

ELIGIBILITY:
Inclusion criteria for sporadic ICA cases:

* Any adult patient consulting for a definite and typical bifurcation AIC authenticated on MRI and/or cerebral arteriography
* Aneurysm discovered less than a year ago, with initial imaging (MRI and/or CTA and DSA) available
* Written consent obtained for study participation
* Patient covered by a social security plan

Inclusion criteria for index and related cases (familial forms) of intracranial aneurysms (ICA):

* Index case: Any adult patient consulting for a definite and typical bifurcation ICA presenting at least one other case with ICA related to the 1st or 2nd degree (child, parent, brother, sister) detected by MRI with at least one Time of Flight (TOF) sequence.
* Family relatives: All 1st- and 2nd-degree relatives (children, parents, brothers, sisters), of legal age, of patients with a family history of definite, typical bifurcation AIC (≥ 2 affected), Screening to be performed using MRI with at least a Time of Flight (TOF) sequence.
* Written consent to participate in the study
* Patient and relatives covered by a social security plan

Exclusion Criteria:

* Syndromic diagnosis known to cause ICA: Marfan syndrome, OSA with SMAD 3, Elhers Danlos syndrome type II and IV, Autosomal Dominant Cystic Fibrosis, Moya-Moya syndrome
* AIC with : Dissecting or fusiform, Associated with arteriovenous malformation, Blister-like, Mycotic
* Cerebral white matter pathology detected on MRI evoking : Col4a1 mutation
* Patient under guardianship or conservatorship
* Person under court protection
* Contraindication to an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Performance of a predictive model allowing the classification of ICA subphenotypes | 36 months
  The performance of a predictive model allowing the classification of ICA subphenotypes will be analysed through the study of genetic results, quantitative features extracted from imaging and clinical data on rupture

SECONDARY OUTCOMES:
Characterization of arterial bifurcations | 36 months
  Quantitative morphological measurements of arterial bifurcations assessed using image processing tools enabling automatic characterization (artery diameters (in mm); artery cross-sections (in mm²); angles separating arteries (in degrees)
Characterization of aneurysmal sacs | 36 months
  Quantitative morphological measurements of aneurysmal sacs assessed using image processing tools enabling automatic characterization (volume (in mm³); external surface area of the envelope (mm²); neck area (mm²))
Screening of genetic mutations | 36 months
  Presence of genetic mutations in patients with intracranial aneurysms compared with a reference population, but also in a familial context. Genetic variations will be studied by whole exome sequencing
Correlation between genotypes and phenotypes | 36 months
  Correlations between genetic mutations and the different clinical and biological phenotypes described in patients with sporadic ICA

CONTACTS AND LOCATIONS:
Overall Officials: Romain BOURCIER, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided